CLINICAL TRIAL: NCT02859389
Title: Neurocognitive and Psychosocial Outcomes in Survivors of Childhood Leukemia With Down Syndrome
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DSCOG
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2018-09

CONDITIONS: Leukemia; Down Syndrome
Keywords: Leukemia; Down Syndrome; Neurocognitive; Survivorship; Attention; Executive function; Late effects
MeSH Terms: conditions — Leukemia; Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survivors of acute lymphoblastic leukemia (ALL) are at risk for neurocognitive deficits, reduced educational and psychosocial outcomes, and lower quality of life. Neurocognitive assessment is frequently implemented during therapy and continued into survivorship to monitor functioning and to facilitate intervention. Children with Down Syndrome (DS) are at 10 to 20-fold increased risk for leukemia. Survival rates for leukemia patients with DS are comparable to or lower than patients without DS, however, these patients are at greater risk for treatment-related toxicities. Children with preexisting neurodevelopmental conditions, including DS, are systematically excluded from neurocognitive assessment on clinical trials, contributing to a gap in the investigators understanding of outcomes in these patients with preexisting neurocognitive vulnerability. The investigators propose a novel preliminary investigation of functional outcomes in children with DS and childhood leukemia. This study has implications for future treatment of leukemia patients with DS, and may generalize to leukemia patients with other predispositions or preexisting neurodevelopmental conditions (e.g., genetic disorders, acquired brain injury, autism, and epilepsy).

Primary Objective:

* To describe neurocognitive and psychosocial outcomes in survivors of childhood leukemia with Down Syndrome using a novel assessment approach.

DETAILED DESCRIPTION:
The investigators will recruit survivors of childhood leukemia with DS to participate in a one-time assessment of neurocognitive and psychosocial functioning. Potentially eligible families will be identified via medical record review at St. Jude Children's Research Hospital (SJCRH) and contacted to discuss study objectives, assess interest, and confirm eligibility. Eligible families will be scheduled for one study visit, estimated to last about 2.5 hours. Participants will provide informed consent prior to the start of any study procedures. Survivors who are ≥ 5 years old will complete performance-based neurocognitive measures. Caregivers (i.e., parents or legal guardians) of all participants, regardless of age, will complete ratings of executive function, behavior, and adaptive skills. Participants will be asked to identify and provide written permission to contact a secondary informant (e.g., teacher or work supervisor). Identified informants will be contacted by study team members and asked to complete behavior rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an SJCRH patient with a diagnosis of leukemia.
* Diagnosis of Trisomy 21 DS as documented in the medical record
* Completed all cancer-directed therapy at SJCRH, since 1980, and at least 6 months prior to the study visit
* English as the primary language

Exclusion Criteria:

* Documented history of central nervous system (CNS) injury or disease that occurred after completing cancer-directed therapy
* History of or current substance use or abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have Down Syndrome and will have been treated for childhood leukemia at St. Jude Children's Research Hospital (SJCRH).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Outcome | Once at participant enrollment
  Descriptive statistics will be estimated.
Psychosocial Outcome | Once at participant enrollment
  Descriptive statistics will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Jacola, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols